CLINICAL TRIAL: NCT07281456
Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Primary Sjogren s Disease Phase IIa Open-Label Placebo-Controlled Clinical Trial and Associated Mechanistic Studies
Brief Title: Safety of Tofacitinib, an Oral Janus Kinase Inhibitor, in Primary Sjogren Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002290; 002290-D
Record Dates: First submitted 2025-12-12; First posted 2025-12-15 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12-29

CONDITIONS: Sjogren's Syndrome
Keywords: Salivary; Dry Mouth; Safety; Inflammation; Xerostomia; Jak; Autoimmune; Xerophthalmia; Lacrimal; Exocrine
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Inflammation; Xerophthalmia | interventions — tofacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug: Tofacitinib (Experimental): Sjogren's Disease (SjD) patients with mild to moderate disease activity receive tofacitinib 5 mg orally twice daily for 168 days.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — XELJANZ(R) is the citrate salt of tofacitinib. Tofacitinib citrate is a white to off-white powder. XELJANZ(R) is supplied for oral administration as 5 mg tofacitinib (equivalent to 8 mg tofacitinib citrate) white round, immediate-release film-coated tablet.

SUMMARY:
Background:

Sjogren disease is an autoimmune disease - that is, a disease that causes the body's immune system to attack its own organs and tissues. Sjogren disease can affect the kidneys, lungs, or other organs. It can also cause dry mouth and eyes, fever, joint pain, rashes, and other symptoms. Researchers want to know if a drug approved to treat rheumatoid arthritis and other autoimmune diseases can help people with Sjogren disease.

Objective:

To test a drug (tofacitinib) in people with Sjogren disease.

Eligibility:

People aged 18 to 75 years with Sjogren disease. They must be enrolled in protocol 15-D-0051.

Design:

* Participants will be screened. They will have a physical exam with blood and urine tests. They will give samples of saliva; a small sample of tissue will be taken from a salivary gland. They will have a test of their heart function. They will have an eye exam, including a test for dry eyes.
* Tofacitinib is a tablet taken by mouth. Participants will take the drug twice a day at home.
* Participants will have 9 clinic visits over 28 weeks. Each visit will take up to 5 hours. In addition to repeated tests, they will have tests of the speed and pressure of blood flow through their body. They will complete health questionnaires throughout the study.
* Participants will also have 5 phone visits during the study. They will review their health and study treatments.
* They will have 1 final visit after they stop taking the drug.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

As a primary objective, this study represents an innovative investigative measure of the safety and tolerability of JAK inhibition in participants with Sjogren's disease. Secondary objectives will include investigating the effects of Tofacitinib on target tissues (e.g., salivary gland function), systemic inflammation, and on vascular function in SjD participants. We also aim to identify biomarkers of response that may be useful as endpoints in future studies.

OBJECTIVES:

Primary Objective:

-To determine the safety and tolerability of Tofacitinib in participants with SjD and mild to moderate disease activity.

Secondary Objectives:

* To assess clinical improvement after treatment with Tofacitinib as measured by changes in the European League Against Rheumatism (EULAR) Sjogren's Disease Activity Index (ESSDAI) and no worsening on the Physician's Global assessment Scale (PGA).
* To demonstrate that treatment with Tofacitinib is effective clinically and biologically in SjD individuals with mild to moderate disease.
* To investigate the effects of Tofacitinib on systemic biomarkers of SjD as measures biological effects that can be used as outcome measures to power a larger Clinical Trial.

ENDPOINTS:

Primary Endpoint:

-Safety and tolerability will be measured by assessment of adverse events (AEs) and clinical safety laboratory tests throughout the study. Toxicity is defined as any Tofacitinib-related Grade 3 adverse event or higher (as measured by the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0) and number and rates of SjD disease flares.

Secondary Endpoints:

Preliminary assessments of clinical response will be measured by:

* Changes in the ESSDAI score between Baseline and Day 168 (end of treatment)
* Changes in the Physician's Global Assessment (PGA) scores between baseline and study day 168.
* Changes in serum cytokines, autoantibody levels (e.g., ANAHep2 substrate, SSA, SSB autoantibody titers), complement proteins C3 and C4, markers of systemic inflammation such as ESR and CRP between baseline and study day 168

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult SjD participants with mild-to-moderate disease activity will be eligible for this study. Enrolled participants can be naive or failed immunosuppressive therapy beyond antimalarials and glucocorticoids; to prevent bias in the cohort of participants with more recalcitrant disease. We expect that Tofacitinib is a potential second line therapy, in addition to antimalarials and glucocorticoids, depending on the participant's initial presentation and response. Women and members of minority groups, if eligible, will be included in accordance with the NIH Policy on Inclusion of Women and Minorities as Participants in Research Involving Human Participants.

Additionally, 20-D-0131(Safety of Tofacitinib, an oral Janus Kinase Inhibitor, in primary Sjogren's syndrome Phase Ib-IIa placebo-controlled clinical trial and associated mechanistic studies) participants who at unblinding received placebo will be contacted and asked to return to the study to participate in this study.

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability of participant to understand and the willingness to sign a written informed consent document.
2. Participation and enrollment in companion protocol, 15-D-0051, Characterization of Diseases with Salivary Gland Involvement.
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Male or female, aged between 18-75 years
5. In good general health as evidenced by medical history
6. Meets the 2002 American European Consensus Group classification criteria for Sjogren's disease or 2016 American College of Rheumatology/European League against Rheumatism Classification Criteria (ACR-EULAR) with mild to moderate disease activity defined as ESSDAI between 0 to 13 at the screening visit and >0 ml/min/gland stimulated saliva flow.
7. Ability to take oral medication and be willing to adhere to the study intervention regimen
8. If on glucocorticoids, the dose must be less than 10 mg daily and stable for the 4 weeks (28 days) prior to screening visit.
9. If on hydroxychloroquine or other antimalarials such as chloroquine or quinacrine, the dose must have been stable for the 12 weeks (96 days) prior to screening visit. The maximum allowed dose is hydroxychloroquine up to 400 mg/day or 6.5 mg/kg/day if more than 400 mg/day. The maximum allowed dose for chloroquine phosphate is up to 500 mg daily and for quinacrine up to 100 mg daily.
10. Participants may be on lipid lowering medications if initiated at least 3 months prior to the screening visit and dose must be stable for 4 weeks (28 days) prior to study entry.
11. Males and females with potential for reproduction must agree to practice effective birth control measures. Females should be on adequate contraception if they are of child-bearing potential documented by a clinician, unless participants or spouse have previously undergone a sterilization procedure. Adequate birth control measures are: intrauterine device (IUD) alone or hormone implants, hormone patches, injectable, or oral contraceptives plus a barrier method (male condom, female condom or diaphragm), abstinence or a vasectomized partner.
12. Agreement to adhere to Lifestyle Considerations throughout study duration

EXCLUSION CRITERIA:

To be eligible to participate in this study, an individual must not meet any of the following criteria:

1. Current or prior treatment with rituximab, belimumab, or any other biologic agent in the 6 months prior to screening.
2. Current or prior treatment with Tofacitinib for more than 6 months in the last 2 years prior to screening.
3. Current treatment with methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus, or other less common immunomodulatory drugs such as those falling into the class of disease-modifying antirheumatic drugs (DMARDs), not otherwise specified herein. Participants previously on methotrexate, azathioprine, mycophenolate mofetil, cyclosporine or tacrolimus, or other DMARDs should have withdrawn drug for at least 8 weeks (56 days) at the time of screening. The use of topical or ophthalmic preparations of cyclosporine, tacrolimus, or other DMARDs is permitted and does not require an 8-week withdrawal period.
4. Treatment with cyclophosphamide, pulse methylprednisolone or IVIG within 6 months prior to screening.
5. Current treatment with potent inhibitors of Cytochrome P450 3A4 (CYP3A4) (e.g., ketoconazole) or receiving one or more concomitant medications that result in both moderate inhibition of CYP3A4 and potent inhibition of CYP2C19 (e.g., fluconazole) that would increase serum availability of Tofacitinib. Past treatment with the agent is allowed if it was more than a week prior to the administration of the first dose of study medication.
6. History of chronic liver disease, not including well-controlled Sjogren's-related chronic liver disease or elevated LFTs:

   * ALT or AST >= 2x upper limit of normal at screening
   * Serum unconjugated bilirubin > 2mg/dL at screening
7. Serum creatinine >1.5mg/dL.
8. Protein to creatinine ratio of more than 1mg/dL at screening (repeated and confirmed three times or confirmed with 24 hours urine protein of more than 1000mg).
9. Active urinary sediment (WBC, RBC or mixed cellular casts 1+ or more /hpf).
10. Hypercholesterolemia: Values after 8-12 hour fasting blood specimen: total cholesterol >250 mg/dL or LDL >180 mg/dL or hypertriglyceridemia (triglyceride >300 mg/dL) within - 45 days of screening visit.
11. WBC <2500/microL or ANC <1,000/microL, Hgb <9.0 g/dL or platelets <70,000/microL or absolute lymphocyte count < 500/microL.
12. Pregnant or lactating women. Women of childbearing potential are required to have a negative pregnancy test at screening.
13. A history of drug or alcohol abuse within the 6 months prior to screening.
14. Currently receiving hemodialysis, peritoneal dialysis, or intestinal dialysis.
15. Active infection that requires the use of oral or intravenous antibiotics unresolved at least 14 days prior to the administration of the first dose of study medication.
16. Active chronic infections including but not limited to HIV, Hepatitis B, Hepatitis C, and BK viremia at screening visit.
17. Current or previous diagnosis of malignant disease, except for basal cell or squamous cell carcinoma of the skin with complete excision and clear borders or adequately treated in situ carcinoma of the cervix.
18. Known active tuberculosis. Participants with treated latent tuberculosis (LTB) will be eligible to participate. Participants with untreated LTB will not be excluded but will be evaluated by an infectious disease (I.D.) consultant and may become eligible for trial based on infectious disease consultant recommendations.
19. History of severe or systemic infections caused by common pathogens, or history of infection with pathogens that do not normally cause human disease.
20. Participants with active renal or central nervous system disease or a high activity level in any organ system (except articular) in ESSDAI54.
21. Participants with known increased risk factors for major adverse cardiac event (MACE) including a history of:

    * Ischemic heart disease (e.g., history of acute myocardial infarction)
    * Heart failure
    * Cardiomyopathy
    * Severe valvular heart disease
    * Significant arrhythmias
    * Chronic renal failure
    * Cerebrovascular accident or transient ischemic attack
    * Uncontrolled diabetes mellitus
    * Uncontrolled hypertension
    * Current smokers or former smokers with less than 3 years since complete cessation and/or >20 pack-years of smoking history.
22. Significant impairment of major organ function (lung, heart, liver, kidney) or any condition that, in the opinion of the Investigator, would jeopardize the participant's safety following exposure to the Tofacitinib.
23. Known history of arterial or venous thrombosis or at high risk for clotting disorder
24. Psychiatric illness or history of medical non-compliance that the study team feels will make the patient unlikely to complete the study
25. Uncontrolled thyroid disease as determined by PI or medically responsible investigator.
26. Known allergic reactions to Tofacitinib or its components
27. Treatment with another investigational drug/intervention within six months except for COVID-19 vaccines or therapies that have been granted an FDA emergency authorization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2030-12-15 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events by Grade/Category | Up to Day 196
  Count of adverse events by grade was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to adverse event. Serious is defined as any grade 3 or higher adverse event. Toxicity is defined as any study drug-related Grade 3 or higher adverse event.
Participants With Adverse Events | Up to Day 196
  Number participants with any adverse events by grade and severity was assessed using the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activity of daily living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event. Serious is defined as any grade 3 or higher adverse event. Toxicity is defined as any study drug-related Grade 3 or higher adverse event.

SECONDARY OUTCOMES:
Change in Physicians Global Assessment (PGA) Score | Day 168 minus Day 1
  The Physician Global Activity (PGA) is a subjective physician reported disease activity index that uses a 10-cm Visual Analog Scale (VAS) to score a patient's disease activity. The 10-cm visual analogue scale (VAS) was scored by a physician with a vertical line on the scale marking disease activity where 0 cm indicates no evidence of disease activity, and 10 cm indicates severe disease activity, with score reported on a scale from 0-10. Higher score indicates more disease activity. Change in disease activity index was measured as the mean difference in disease activity scores between time points. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Change in EULAR Sj(SqrRoot)(Delta)gren's Syndrome (SS) Disease Activity Index (ESSDAI) Score | Day 168 minus Day 1
  The EULAR Sjogren's syndrome (SS) disease activity index (ESSDAI) is a systemic disease activity index designed to measure disease activity in patients with primary SS. It includes 12 organ domains (e.g., constitutional, glandular, neurological) for disease activity, each with a 4-point scale (0 = No activity; 3=High activity). These scores are then multiplied by domain-specific weights (1-6) and summed to produce a total score ranging from 0 to 123, with higher scores indicating greater disease activity. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Change in Whole Unstimulated Saliva Flow | Day 168 minus Day 1
  Changes in salivary flow was assessed by measuring whole unstimulated saliva flow (WUS) and glandular parotid and submandibular/sublingual unstimulated and 0.2% citric acid stimulated flow rates using ultrasonograph. Validated scoring criteria was used to assess ultrasonographic feature parameters at baseline and at the study day 168. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Change in Whole Stimulated Saliva Flow | Day 168 minus Day 1
  Changes in salivary flow was assessed by measuring whole stimulated saliva flow and glandular parotid and submandibular/sublingual stimulated and 0.2% citric acid stimulated flow rates using ultrasonograph. Validated scoring criteria was used to assess ultrasonographic feature parameters at baseline and at the study day 168. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.
Change in EULAR Sj(SqrRoot)(Delta)gren's Syndrome (SS) Patient Reported Index (ESSPRI) | Day 168 minus Day 1
  The EULAR Sjogren's Syndrome (SS) Patient Reported Index (ESSPRI) is a patient-reported outcome measure (PROM) that focuses on the subjective experience of symptoms in SS. The tool assesses the key symptoms of dryness, pain and fatigue. A single 0-10 numerical scale is used to assess each of these symptoms. Final score is the average of the scores from the three domains. A final ESSPRI score of less than 5 is considered indicative of acceptable disease status, while a score of 5 or higher suggests high disease activity. Questionnaire was completed at baseline and day 168. Data was analyzed as the change in score between day 1 (baseline) and study day 168 (Change = day 168 - day 1) for the treatment/placebo groups as repeated measures.

CONTACTS AND LOCATIONS:
Overall Officials: Blake M Warner, D.D.S., Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Study complies with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule.
Time Frame: At the time of publication or after 3 years, whichever comes first.
Access Criteria: This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002290-D.html